CLINICAL TRIAL: NCT01093664
Title: Phase IB Follow-up Study to Assess a Boost Immunization With AFFITOPE AD02 With Regard to Safety/Tolerability, Immunological and Clinical Activity in Alzheimer Patients Who Have Received the Vaccine Within the Clinical Study AFF002
Brief Title: Safety/Tolerability, Immunological and Clinical Activity of a Boost Immunization With AFFITOPE AD02
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Affiris AG (Industry)
Responsible Party: Achim Schneeberger, MD, AFFiRiS AG
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFF004A
Record Dates: First submitted 2009-09-02; First posted 2010-03-26 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AFFITOPE AD02 (Experimental)
  Interventions: Biological: AFFITOPE AD02

INTERVENTIONS:
Biological: AFFITOPE AD02 — s.c. injection

SUMMARY:
This is a phase IB follow-up study to assess a boost immunization with AFFITOPE AD02 with regard to safety/tolerability, immunological and clinical activity in Alzheimer patients who have received the vaccine within the clinical study AFF002.

ELIGIBILITY:
Inclusion Criteria:

* Participation in AFF002 and AFF004

Exclusion Criteria:

* Presence or history of allergy to components of the vaccine, if considered relevant by the investigator
* Contraindication for MRI imaging
* History and/or presence of autoimmune disease, if considered relevant by the investigator
* Active infectious disease (e.g., Hepatitis B, C)
* Presence and/or history of Immunodeficiency (e.g., HIV)
* Significant systemic illness

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | July 2010
  * Withdrawal criteria (continuation decision) Number of patients who withdraw due to AEs Reason for withdrawal
  * Adverse events (AEs)
  * Serious adverse events (SAEs)
  * Physical and neurological examination
  * Concomitant medication
  * Vital signs (blood pressure, heart rate, respiratory rate, body temperature)
  * Body mass (weight and height)
  * MRI of brain
  * ECG
  * Laboratory assessment (haematology, biochemistry, coagulation, serology and urinalysis)

SECONDARY OUTCOMES:
Immunological and clinical activity | July 2010
  Immunological parameters:
  - Assessment of the immune response triggered by the vaccine (titre of IgG antibodies specific for the immunizing peptide, N-terminal part of Aβ, (irrelevant peptide serves as specificity control), Aβ itself and KLH as assessed by ELlSA as well as the results of the biacore affinity measurements towards the immunizing peptide and Aβ)
  Clinical efficacy variables:
  * Cognitive and functional tests, behavioural scales
  * Measurement of quality of life in patients with Alzheimer's disease
  * Investigator's global evaluation scale

CONTACTS AND LOCATIONS:
Overall Officials: Margot Schmitz, Univ. Doz., Principal Investigator — Ordination Schmitz
Locations (1):
- Ordination Schmitz, Vienna, Vienna, Austria